CLINICAL TRIAL: NCT04323735
Title: Intravesical Lactobacillus for Urinary Symptoms Among People With NLUTD Who Use Indwelling Catheters
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Children's National Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001782
Record Dates: First submitted 2020-01-28; First posted 2020-03-26 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Neurogenic Bladder
Keywords: Indwelling catheter; Foley catheter; Suprapubic Catheter
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Design: Prospective, randomized pilot intervention clinical trial. Target Enrollment: 182 subjects with NLUTD at least 6 months and who use IDC for bladder management. Setting: National sample (N=114 intervention only, no urine collection) and local Washington, DC metropolitan area (N=68 intervention + urine collection).
  Controls: This is a 2-arm dose-finding pilot clinical trial, as such there is no control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dosage (Active Comparator): For the LGG® instillation, participants will be instructed to mix the contents of 1 LGG capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG mixture into a 60cc syringe and instill via the indwelling catheter (the catheter will not be changed as this would represent 2 interventions). Participants will be instructed the plug their catheter for 1 hour. Participants will receive 2 ]LGG capsules and will repeat this process the following day ("Low" dose). Subjects will remain in the study for up to 29 months, with participation ending after one completed intervention (2 doses) and post-intervention assessments are complete. If urinary symptoms do not occur warranting instillation during the ensuing 29 months, participants will be asked to return any remaining kits (including LGG®). Participants will be instructed to complete the USQNB-IDC weekly until study completion.
  Interventions: Drug: Culturelle 10 Billion CFU Capsule
- High dosage (Active Comparator): For the LGG® instillation, participants will be instructed to mix the contents of 1 LGG capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG mixture into a 60cc syringe and instill via the indwelling catheter (the catheter will not be changed as this would represent 2 interventions). Participants will be instructed the plug their catheter for 1 hour. Participants will receive 4 LGG capsules and will repeat this process the following day twice for a total of four doses ("High" dose). Subjects will remain in the study for up to 29 months, with participation ending after one completed intervention (4 doses) and post-intervention assessments are complete. If urinary symptoms do not occur warranting instillation during the ensuing 29 months, participants will be asked to return any remaining kits (including LGG®). Participants will be instructed to complete the USQNB-IDC weekly until study completion.
  Interventions: Drug: Culturelle 10 Billion CFU Capsule

INTERVENTIONS:
Drug: Culturelle 10 Billion CFU Capsule — LGG® (Culturelle Probiotic with Lactobacillus RhamnosusGG, shown to produce the largest amount of antibacterial substances against pathogenic bacteria) will be used. For the LGG® instillation, participants will be instructed to mix the contents of 1 LGG capsule into 45 cc sterile 0.9% saline. After mixing, participants will draw up the 45cc liquid LGG mixture into a 60cc syringe and instill via the indwelling catheter (the catheter will not be changed as this would represent 2 interventions). Participants will be instructed the plug their catheter for 1 hour. Participants will receive 2 or 4 LGG capsules (depending on randomization group) and will repeat this process the following day ("Low" dose) or twice daily for a total of four doses ("High" dose) according to randomization group.
  Other Names: Lactobacillus Rhamnosus GG

SUMMARY:
The objectives of the proposed research among this population are: 1) to define clinically meaningful change (i.e. differentiating states of health and illness) with respect to urinary symptoms, urine inflammation, cultivable bacteria, and the urine ecosystem; and 2) to determine the optimal intravesical Lactobacillus RhamnosusGG (LGG®) dose to be used to reduce urinary symptoms in a future clinical trial.

DETAILED DESCRIPTION:
Urinary tract infection (UTI) is the most common outpatient infection world-wide, and for people with spinal cord injury (SCI) and neurogenic bladder (NB), it is the most common infection, secondary condition, cause for emergency room visits, and infectious cause of hospitalization. Despite its prevalence, attempts to ameliorate UTI among people with SCI are stymied by long-standing diagnostic challenges which arise from evidence gaps around "gold standard" diagnostic tests (urinalysis and urine culture) that have lower sensitivity and specificity for UTI in this population. A high prevalence of chronic inflammation leading to persistence of white blood cells (WBC) in the urine confounds the utility of WBC count, pyuria, and leukocyte esterase as biomarkers for UTI; nitrites in urine indicate the presence of only specific (but not all) organisms, many of which are present to a greater extent in the urine of people with SCI; and people with SCI have a high prevalence of asymptomatic bacteriuria. These physiologic changes render the gold standard diagnostic tests less useful for identifying UTI in persons with SCI.

SA1. Estimate healthy, asymptomatic state variability of urine NGAL (uNGAL), white blood cells (uWBC), nitrite, cultivable bacteria, and the urinary microbiome.

SA2. Estimate the effect of intravesical LGG dose on urinary symptoms (primary outcome), uNGAL, uWBC, nitrites, cultivable bacteria, and the urine microbiome (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Neurogenic bladder for at least 6 months;
* Utilizing indwelling catheterization for bladder management;
* Women must be premenopausal and not currently menstruating;
* Community dwelling
* physical disability

Exclusion Criteria:

* Use of prophylactic antibiotics;
* Instillation of intravesical antimicrobials to prevent UTI;
* Psychologic or psychiatric conditions influencing the ability to follow instructions;
* Use of oral or IV antibiotics within the past 2 weeks;
* Sexual activity within the previous 72 hours;
* Participation in another study with which results could be confounded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 1) day of urine collection
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes. (local urine collection participants only)
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 1) day 1 post urine collection
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes. (local urine collection participants only)
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 1) day 2 post urine collection
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes. (local urine collection participants only)
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 1) day 3 post urine collection
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes. (local urine collection participants only)
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) Weekly up to 29 months
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) day 1 of intervention (low or high dose)
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes. (local urine collection participants only)
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) day 2 of intervention (low or high dose)
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) day 3 of intervention (low or high dose)
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) day 4 of intervention (low or high dose)
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) day 5 of intervention (high dose only)
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes
Urinary Symptom Questionnaire for Neurogenic Bladder- Indwelling catheter | (SA 2) 24-48 hours after intervention completion
  Will measure change in urinary symptoms for those that use an indwelling catheter. Higher score may mean worse outcomes. (local urine collection participants only)
Change in Urine white blood cell count | (SA 1) day 1 post urine collection
  urinalysis. (local urine collection participants only)
Change in Urine white blood cell count | (SA 1) day 14 post urine collection
  urinalysis. (local urine collection participants only)
Change in Urine white blood cell count | (SA 2) day 1 of intervention
  urinalysis. (local urine collection participants only)
Change in Urine white blood cell count | (SA 2) 24-48 hours after intervention completion
  urinalysis. (local urine collection participants only)
Change in Urine Nitrite | (SA 1) day 1 post urine collection
  urinalysis. (local urine collection participants only)
Change in Urine Nitrite | (SA 1) day 14 post urine collection
  urinalysis. (local urine collection participants only)
Change in Urine Nitrite | (SA 2) day 1 of intervention
  urinalysis. (local urine collection participants only)
Change in Urine Nitrite | (SA 2) 24-48 hours after intervention completion
  urinalysis. (local urine collection participants only)
Change in Urine NGAL | (SA 1) day 1 post urine collection
  Urine NGAL. (local urine collection participants only)
Change in Urine NGAL | (SA 1) day 14 post urine collection
  Urine NGAL. (local urine collection participants only)
Change in Urine NGAL | (SA 2) day 1 of intervention
  Urine NGAL. (local urine collection participants only)
Change in Urine NGAL | (SA 2) 24-48 hours after intervention completion
  Urine NGAL. (local urine collection participants only)
Change in Cultivable Bacteria | (SA 1) day 1 post urine collection
  urine culture. (local urine collection participants only)
Change in Cultivable Bacteria | (SA 1) day 14 post urine collection
  urine culture. (local urine collection participants only)
Change in Cultivable Bacteria | (SA 2) day 1 of intervention
  urine culture. (local urine collection participants only)
Change in Cultivable Bacteria | (SA 2) 24-48 hours after intervention completion
  urine culture. (local urine collection participants only)
Change in Urine microbiome composition and function | (SA 1) day 1 post urine collection
  Next generation sequencing for microbiome composition. (local urine collection participants only)
Change in Urine microbiome composition and function | (SA 1) day 14 post urine collection
  Next generation sequencing for microbiome composition. (local urine collection participants only)
Change in Urine microbiome composition and function | (SA 2) day 1 of intervention
  Next generation sequencing for microbiome composition. (local urine collection participants only)
Change in Urine microbiome composition and function | (SA 2) 24-48 hours after intervention completion
  Next generation sequencing for microbiome composition. (local urine collection participants only)
NINDS Medical History CDE: | Baseline
  A brief medical history using body system categories
Medical History Form | Baseline
  Medical history of participant
International SCI Lower Urinary Tract Function Basic Data Set | Baseline
  A tool to describe urinary tract impairment, awareness of need to empty the bladder, main bladder emptying method, medications used for bladder management, surgeries, and change in urinary symptoms in the past year.
NINDS Prior and Concomitant Medications CDE | Baseline
  Contains whether or not the participant is taking a medication during the study protocol, name of medication, reason for medication, medication dose, frequency, start and end dates, and free text

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Groah, MD, MSPH, Principal Investigator — MedStar National Rehabilitation Hospital
Locations (1):
- MedStar National Rehabilitation Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No